## **Title Page**

**Type of Article:** Prospective Observational

**Manuscript Title:** Effect of Respiratory Exerciser on Pulmonary Functions of COVID-19 patients; A Prospective Observational Study

Running Head: Respiratory Exerciser on COVID-19

**Document Date:** 08.02.2021

**NCT Number:** 04826731

## **Authors**

Yasemin Aydın<sup>1</sup>, Emergency Medicine Specialist, MD, ysmnyaydin@gmail.com, ORCID:

Aynur Yurtseven<sup>1</sup>, Emergency Medicine Specialist, MD, aynuryurt7@gmail.com, ORCID: 0000-0002-1554-0873

Kerem Ensarioğlu<sup>2</sup>, Pulmonary Medicine Resident, MD, kerem.ensarioglu@gmail.com, ORCID: 0000-0002-0968-1549

Bahar Kurt<sup>2</sup>, Pulmonary Medicine Specialist, Professor, MD, baharkurt@yahoo.com, ORCID: 0000-0002-3495-2339

<sup>1</sup>Emergency Medicine Department, Faculty of Health Sciences Dışkapı Yıldırım Beyazıt Training and Research Hospital, Ankara, Turkey

<sup>2</sup>Pulmonary Medicine Department, Faculty of Health Sciences Dışkapı Yıldırım Beyazıt Training and Research Hospital, Ankara, Turkey

## INFORMED CONSENT AND VOLUNTEER INFORMATION FORM

We are conducting a new study on the disease COVID-19. The name of the study is "Evaluation of Lung Capacity after Triflow Use in Patients With COVID-19 Infection and Lung Involvement".

We encourage you to participate in this research as well. However, let's say right away that you are free to participate or not to participate in this research. Participation in the study is on a voluntary basis. We would like to inform you about the research before your decision. If you want to participate in the research after reading and understanding this information, please sign the form.

The reason we want to do this research is to investigate the effect of COVID-19 disease on lung function at follow-up. Your participation in this study, which will be carried out with the joint participation of Health Sciences University Dışkapı Yıldırım Beyazıt Training and Research Hospital Health Application and Research Center Emergency Service and Chest Diseases Clinics, is important for the success of the research.

In order to be accepted into the study, your nasopharyngeal COVID-19 test must be positive. If you are diagnosed with COVID-19 by any other method (such as CT scan and blood antibody test), you will not be considered eligible even though you are evaluated for the study. Another necessary condition for your acceptance to work is that your hospitalization is required and this hospitalization is made to the COVID-19 service. You will also not be included in the study if a place is not available for you in the hospital or hospitalization is not required.

There will be no additional testing from you for the study. The results of routine respiratory tests performed after COVID-19 infection and your general information (age, gender, comorbidities, length of stay, summaries of treatment used) will be evaluated by accessing hospital records.

You will not be charged any fee for your participation in this study. No additional payment will be made to you for participating in the study.

Medical information about you will be kept confidential, but may be reviewed, if necessary, by the officials controlling the quality of the study, ethical committees or official authorities.

You may refuse to participate in this study. Participation in this research is completely voluntary and if you refuse, there will be no change in the treatment applied to you. You also have the right to withdraw your consent at any stage of the study.

## **Statement of Participant**

It was stated to me that a medical research would be conducted at Dışkapı Yıldırım Beyazıt E.A.H Emergency Service and Chest Diseases Clinics, and the above information about this research was conveyed to me. After this information, I was invited to such research as a "participant".

If I participate in this research, I believe that the confidentiality of my information, which should be kept between me and the physician, will be treated with great care and respect during this research. I have been given sufficient confidence that my personal information will be carefully protected during the use of research results for educational and scientific purposes.

I can withdraw from the research without giving any reason during the execution of the project. (However, I am aware that it would be appropriate to notify the researcher in advance that I will withdraw from the research in order not to put the researchers in a difficult situation) Also, I can be excluded from the research by the researcher, provided that no harm is done to my medical condition.

I do not take any financial responsibility for the expenses to be made for the research. I will not be paid either.

I know that the study does not require any additional treatment changes or examinations. I was informed and assured that my participation in the study would not change the treatment given to me in any way. I was informed that I would not be under any financial burden regarding the routine treatment and interventions given to me.

I am not obligated to participate in this research and may not. I have not encountered any compelling behavior regarding my participation in the research. I also know that if I refuse to participate, it will not harm my medical care and my relationship with my physician.

I have fully understood all the explanations given to me. After a certain period of reflection on my own, I decided to take part in this research project as a "participant". I accept this invitation.

A copy of this signed form paper will be given to me.

| Participant |
|----------------------------------------|
| Name and surname: |
| Address: |
| Phone. |
| Signature |
| Physician interviewing the participant |
| Name, surname, title: |
| Address: |
| Phone. |
| Signature |